CLINICAL TRIAL: NCT05076864
Title: Levosimendans Pharmacokinetics in Intensive Care Patients
Brief Title: Levosimendans Pharmacokinetics in Intensive Care Patients. An Observational Study.
Acronym: LEFKIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Claire Rimes-Stigare, Senior Consultant, Karolinska University Hospital
Other Study IDs: 4-1951/2021
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Pharmacokinetics; Metabolites; Intensive Care; Renal Failure; Acute Kidney Injury
MeSH Terms: conditions — Renal Insufficiency; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (plasma), Urine, Ultrafiltration fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Evaluation of the pharmacokinetics of levosimendan and its metabolites in intensive care patients with normal, reduced and dialysis supported renal function.

DETAILED DESCRIPTION:
Aims: To gain a better understanding of the pharmacokinetics of Levosimendan in critically ill patients and in particular in those patients with and without renal failure and in those receiving CRRT. This project may give a better basis to determine whether dose monitoring and adjustment of Levosimendan is necessary to avoid toxicity or under treatment. In order to study Levosimendan pharmacokinetics, the Karolinska laboratory has in parallel developed a method for analysis of the substance and its metabolites.

Research questions:

1. To what extent are Levosimendan and its active metabolites dialysable in patients receiving continuous renal replacement therapy.
2. How do the concentrations of Levosimendan and its active metabolites differ in critically ill patients with and without acute renal failure?

Method:

The is a prospective observational study conducted on adult intensive care units at Karolinska University Hospital.

Study Population: Critical care patients who due to clinical need are prescribed Levosimendan by treating physician will be included into one of three groups based on degree of AKI (KDIGO classification) and need for CRRT. This is a non-interventional study.

Number of patients to be included: we intend to include 4-12 patients per group.

Procedure: The decision to prescribe Levosimendan will be made by treating physicians as will decisions regarding dose, dose adjustment and length of treatment.

Screening for inclusion will occur when a decision to prescribe Levosimendan has been made.

Samples of blood, urine and ultrafiltration fluid from the CRRT circuit are to be analysed to determine concentration of Levosimendan and its metabolites. Plasma concentrations will be obtained, before and after the dialysis filter.

Concentration monitoring will occur over a period of up to 6 days, with test taken at 0, 6 and 20 hours after infusion start and after cessation of Levosimendan every two hours for the first 10 hours and there after twice a day for the next 5 days. A maximum of 30 samples (15 in non CRRT patients) of 1-3ml are taken.

Patient groups:

Group 1: Levosimendan + no AKI or KDIGO AKI stage 1. Group 2: Levosimendan + KDIGO AKI stage 2-3, not CRRT Group 3: Levosimendan + KDIGO AKI stage 1-3 with CRRT.

Analysis:

Analysis of the plasma concentration of Levosimendan and its metabolites (OR-1896, OR-1855) is performed at the clinical pharmacology department, Karolinska University Hospital. Reference substances have been provided by Orion Pharma.

Definitions:

Acute Kidney Failure (AKI) is defined according to the KDIGO definition: Creatinine entry from the baseline (percentage increase) and volume of urine production or CRRT treatment.

ELIGIBILITY:
Inclusion Criteria:

° Adult Intensive care patients in whom treating physicians have judged to be in need of Levosimendan treatment.

Exclusion Criteria:

* Patient <18 years of age
* Pregnancy
* Patients receiving Intermittent hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive Care Unit patients in whom the treating physician has decided due to clinical indication to administer levosimendan. Dose and length of treatment decided by treating physician.
  With Group 1: No renal failure or Acute Kidney Injury(AKI)* stage 1. Group 2: AKI stage 2-3, not receiving renal replacement therapy. Group 3: Receiving continuous renal replacement therapy (CRRT)
  *AKI classification system Kidney Disease Improving Global outcomes (KDIGO)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of levosimendan and OR 1896 1855 in plasma | 1-5 days
  Plasma concentrations of levosimendan and its active metabolites afte Levosimendan infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden